CLINICAL TRIAL: NCT05357612
Title: Characterization of the Serotonin 2A Receptor Selective PET Tracer [18F]MH.MZ in Patients With Neurodegenerative Diseases
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Claassen, Assoc Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 212028
Record Dates: First submitted 2022-04-20; First posted 2022-05-03 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Neurodegenerative Diseases; Parkinson Disease; Parkinson Disease Psychosis
MeSH Terms: conditions — Neurodegenerative Diseases; Parkinson Disease | interventions — pimavanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pimavanserin (Experimental)
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — PD related Psychosis

SUMMARY:
It is hypothesize that patients with clinically diagnosed neurodegenerative diseases will have significantly different receptor occupancy of 5HT2A receptors compared to a healthy age/sex-matched control group. This will be tested by measuring 5HT2A receptor density using the PET radioligand (R)-[18F]MH.MZ in both populations.

DETAILED DESCRIPTION:
It is hypothesized that improvement in psychosis symptoms in patients taking pimavanserin will be associated with increased baseline receptor density (Hypothesis 1A), and increased receptor occupancy of 5HT2A receptors following pimavanserin administration (Hypothesis 1B). This will be done by measuring 5HT2A receptor density using the PET radioligand (R)-[18F]MH.MZ within predefined symptom networks for hallucinations, delusions, and sleep. A PET scan will be obtained in PD patients with psychosis at enrollment to measure baseline 5HT2A receptor density and then again after 6 weeks of pimavanserin. The change in binding between baseline and post-drug treatment window will be used to measure 5HT2A receptor occupancy.

It is hypothesize that improvement in psychosis symptoms in patients taking pimavanserin will be associated with increased functional connectivity and cerebral blood flow within predefined symptom networks for hallucinations, delusions, and sleep. This will be tested by obtaining MRI scans assessing resting state functional connectivity and arterial spin labeling in PD patients with psychosis at enrollment (baseline) and then again after 6 weeks of pimavanserin.

It is hypothesized that functional neuroimaging changes in response to pimavanserin will be associated with baseline 5HT2A receptor density and 5HT2A receptor occupancy after pimavanserin administration. To test this hypothesis, the differences in functional neuroimaging measures and PET 5HT2A receptor will be measured in PD psychosis patients off (at baseline) and on Pimavanserin (post-treatment window).

ELIGIBILITY:
Inclusion Criteria:

* Patient arm - clinical diagnosis of Parkinson disease, diffuse Lewy body disease, multiple systems atrophy, Huntington's Disease, Frontotemporal Dementia, and other variants
* Healthy arm - age and gender matched to patient arm
* Psychosis (presence of hallucinations or delusions) starting after the diagnosis of Parkinson's disease, occurring at least weekly for 4 weeks, severe enough to warrant treatment.
* Study partner available for study visits

Exclusion Criteria:

* Prior stroke or other uncontrolled serious neurological or medical illness
* Contra-indication or inability to tolerate MRI scan
* Use of serotonergic medications in the last 6 weeks
* Incapable of providing independent consent.
* Pregnant or breastfeeding women
* psychosis due to a metabolic, toxic, or primary psychiatric disease
* Deemed unable to complete neurocognitive testing
* For PD Participants: current or prior use of pimavanserin
* Use of antipsychotics in the last 2 weeks

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in 5HT2A receptor density measured using the PET radioligand MH.MZ | Baseline and 6 weeks after intervention of Pimavanserin
  Receptor density (Bmax) of 5HT2A receptors measured using the PET radioligand MH.MZ uptake in regions of interest.
Change in 5HT2A receptor binding occupancy measured using the PET radioligand MH.MZ | Baseline and 6 weeks after intervention of Pimavanserin
  Receptor binding occupancy (RO) of 5HT2A receptors measured using the PET radioligand MH.MZ uptake in regions of interest.

SECONDARY OUTCOMES:
Change in psychosis severity | Baseline and 6 weeks after intervention of Pimavanserin
  Change in psychosis severity 6 weeks after starting pimavanserin, as measured by Clinician-Rated Dimensions of Psychosis Symptom Severity (CRD-PSS)18; Domain I (Delusions). Low scores indicate better outcome.
Change in psychosis severity | Baseline and 6 weeks after intervention of Pimavanserin
  Change in psychosis severity 6 weeks after starting pimavanserin, as measured by Clinician-Rated Dimensions of Psychosis Symptom Severity (CRD-PSS)18; Domain II (Hallucinations). Low scores indicate better outcome.
Changes to functional connectivity and ASL bloodflow | Baseline and 6 weeks after intervention of Pimavanserin
  Changes to functional connectivity and ASL bloodflow (mL/g/min) within pre-defined networks for delusions, hallucinations, and sleep after 6 weeks of Pimavanserin.

CONTACTS AND LOCATIONS:
Overall Officials: Ciaran Considine, PhD, Principal Investigator — Vanderbilt University Medical Center; Richard Darby, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided